CLINICAL TRIAL: NCT06565065
Title: Lymphatic Osteopathic Manipulative Treatment Protocol for Healthy Individuals: A Crossover Self-Controlled Clinical Trial
Brief Title: ImmunoBoost: The Lymphatic Osteopathic Manipulative Treatment Protocol Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Collaborators: American Osteopathic Foundation (Unknown)
Responsible Party: Principal Investigator, Brian Loveless, Chief Medical Officer, WesternU Health/ Professor or OMM/MMM WesternU COMP, Western University of Health Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: P24/IRB/002
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: Osteopathic Manipulative Treatment; Lymphatic Pump Treatment; Immune System; OMT; Complete Blood Count; Cytokines
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be directly told of the order of their treatment or workout sessions in an attempt to blind between OMT and sham treatment. Investigators will be blinded to the order in which participants receive their treatment besides the direct treater and the research assistant. Outcome assessors and statisticians will only analyze coded participant data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Order 1 - Day 0: OMT, Week 3: Sham, Week 6: Exercise (Experimental): Osteopathic Manipulative Treatment (OMT)
  followed by a 3-week washout period and then:
  Sham protocol
  followed by a 3-week washout period and then:
  Exercise protocol.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT); Other: Sham Light Touch; Other: Exercise Protocol
- Order 2 - Day 0: Sham, Week 3: OMT, Week 6: Exercise (Experimental): Sham protocol
  followed by a 3-week washout period and then:
  Osteopathic Manipulative Treatment (OMT)
  followed by a 3-week washout period and then:
  Exercise protocol.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT); Other: Sham Light Touch; Other: Exercise Protocol
- Order 3 - Day 0: Exercise, Week 3: OMT, Week 6: Sham (Experimental): Exercise protocol
  followed by a 3-week washout period and then:
  Osteopathic Manipulative Treatment (OMT)
  followed by a 3-week washout period and then:
  Sham protocol.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT); Other: Sham Light Touch; Other: Exercise Protocol

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — A full standardized lymphatic protocol will be performed, including thoracic inlet left and right, thoracoabdominal release, pelvic diaphragm release, pedal pump, splenic pump, and abdominal lymphatic pump. This treatment will be done by systematically working down and back up. The protocol will last a total of 12 minutes for each participant
Other: Sham Light Touch — A full standardized 12-minute session in which treaters will mimic various osteopathic manipulative techniques at specific anatomical locations without applying pressure or manipulation.
Other: Exercise Protocol — A full standardized moderate-intensity physical activity as defined by the Centers for Disease Control (CDC). Target heart rate for moderate-intensity exercise should be between 64 and 76% of maximum heart rate. To estimate age-related heart rate, subjects' age will be subtracted from 220. Then, that number will be multiplied by 75%, which will be standardized across all subjects in the study. Heart rate will be monitored with the use of an attached pulse-ox monitor. Treadmill speed will be adjusted accordingly so that each subject maintains a heart rate of 75% of their maximum heart rate. A brisk walk will be done on a flat treadmill and no incline will be utilized. Subjects will be allowed a minute of warm-up to get to the appropriate pace/target heart rate.

SUMMARY:
The goal of this clinical trial is to determine whether osteopathic manipulative treatment (OMT) enhances immune system readiness in healthy adults compared to exercise or sham light treatment. Specifically, the goal of this study is to assess circulating immune cells and signaling molecules in the blood in response to these various treatments.

It aims to compare: Complete Blood Counts (CBC) and blood immune signaling molecule levels in healthy adults in response to OMT, sham light touch, and exercise, with measurements taken at multiple time points.

Researchers will compare immune blood cells and signaling molecules in response to OMT versus sham light touch and exercise within the same group of healthy adults measured at three time points for each of the three total visits.

Participants will do a 15-minute OMT session, a 15-minute light sham session, or a 15-minute exercise session at each of their three separate visits (they will do one of each over the course of their 3 appointments in random order). They will have three blood draws taken at each of those three visits. They will also fill out a Global Physical Activity Questionnaire (GPAQ) survey to assess their level of physical activity throughout the study.

DETAILED DESCRIPTION:
This clinical trial is a follow-up on a recent trial demonstrating an enhanced immune response in participants who received lymphatic osteopathic manipulative treatment (OMT) with each of their COVID-19 mRNA vaccinations. Similar immune enhancement was observed in a pilot study with OMT in conjunction with the Hepatitis B vaccine. Additionally, animal studies have shown that lymphatic pump OMT can cause transient increases in the movement of lymphatic fluid, immune cells, and signaling molecules throughout the body and bloodstream. These findings were further supported by in vitro studies on fibroblasts, where OMT led to significant increases in circulating cytokines. There are studies that suggest that combining physical exercise with vaccination can also improve immune responses. To parse out these effects observed in OMT and exercise studies and provide the mechanisms underlying the observed immune enhancements, this clinical trial will be conducted.

This study is designed as a crossover, self-controlled, comparative effectiveness randomized clinical trial. A total of 30 healthy individuals who meet all inclusion/exclusion criteria will be recruited. Participants will then fill out a health questionnaire during the screening process to confirm their eligibility.

Each participant will be randomly assigned to one of three intervention sequences to maintain blinding and control for order and sequencing effects. The intervention sequences are as follows:

* Order 1: Day 0: OMT, Week 3: Sham, Week 6: Exercise
* Order 2: Day 0: Sham, Week 3: OMT, Week 6: Exercise
* Order 3: Day 0: Exercise, Week 3: OMT, Week 6: Sham

There will be a 3-week washout period between each intervention. Participants will complete the Global Physical Activity Questionnaire (GPAQ) survey to identify their current level of exercise at each visit. They will also be monitored for any adverse effects following each intervention.

All treatment protocols will be done for a 12-minute timeframe per session. Participants will have three blood draws at each visit: at baseline, five minutes after intervention, and four hours after intervention. The primary outcome measures will include cytokine levels and circulating leukocyte levels, which will be compared across the different intervention sequences.

This study aims to provide a deeper understanding of the mechanism by which lymphatic OMT alters the immune system. It will also compare these effects to the mechanisms of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be 18 years or older.
* Individuals must provide informed consent.
* Individuals must be healthy with a BMI under 30, with no primary or secondary immune deficiency or autoimmune disease/must not be immunocompromised.
* Individuals must not be using or recently have used any immune-altering medications such as corticosteroids, cyclosporin, tacrolimus, and pimecrolimus
* Individuals must not have had lymphatic OMT or other physical manipulation such as acupuncture, physical therapy, chiropractic, or massage therapy in the previous four weeks before study enrollment.
* Individuals must have the ability to receive OMT with lymphatic techniques.
* Individuals must be able to tolerate 12 minutes of moderate physical activity.
* Individuals must not be pregnant or breastfeeding.
* Individuals must not have had a splenectomy or other spleen or oncologic surgery within the past 6 months.
* Individuals must be infection-free for the past 6 weeks before starting the study and have not received any immunizations within the past 6 weeks.
* Individuals must be willing to avoid strenuous activity at least 24 hours before each visit.
* Individuals must be willing to abstain from moderate to intense activity in the 4 hours between their 2nd blood draw and their final blood draw at each of their three visits.

Exclusion Criteria:

* Individuals are younger than 18 years of age.
* Individuals who do not provide informed consent.
* Individuals with a BMI over 30, or with primary or secondary immune deficiency or autoimmune disease or is immunocompromised.
* Individuals using or recently have used any immune-altering medications such as corticosteroids, cyclosporin, tacrolimus, and pimecrolimus
* Individuals who have had lymphatic OMT or other physical manipulation such as acupuncture, physical therapy, chiropractic, or massage therapy in the previous four weeks before study enrollment.
* Individuals who don't have the ability to receive OMT with lymphatic techniques.
* Individuals who cannot tolerate 12 minutes of moderate physical activity.
* Individuals who are pregnant or breastfeeding.
* Individuals who have had a splenectomy or other spleen or oncologic surgery within the past 6 months.
* Individuals who have had an infection in the 6 weeks before starting the study and or have received any immunizations within the past 6 weeks.
* Individuals not willing to avoid strenuous activity at least 24 hours before each visit.
* Individuals not willing to abstain from moderate to intense activity in the 4 hours between their 2nd blood draw and their final blood draw at each of their three visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Complete Blood Count (CBC) with differential | Baseline to 5 minutes post-intervention to 4 hours post-intervention.
  CBC with differential will be evaluated to identify the number of circulating plasma leukocytes for each intervention for each of the three interventions at three time points for each visit/intervention. This test will help us identify levels of erythrocytes, platelets, and leukocytes, including neutrophils, lymphocytes, monocytes, eosinophils, and basophils. This will be compared across time points for OMT, sham treatment, and exercise.

SECONDARY OUTCOMES:
Pro-Inflammatory cytokine profiling | Baseline to 5 minutes post-intervention to 4 hours post-intervention.
  V-Plex Human Proinflammatory Panel I (4-Plex) will be used to identify cytokine profiles, including including IL-6 (Interleukin-6), IL-1β (Interleukin-1 beta), INF-γ (Interferon-gamma), and TNF-α (Tumor Necrosis Factor-alpha). This will be evaluated for each of the three interventions at three time points for each visit/intervention. This will be compared across time points for OMT, sham treatment, and exercise.
Evaluation of safety based on reported adverse events | Through study completion, an average of 6 weeks.
  Documentation of any adverse events to OMT, sham treatment, or exercise protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Loveless, DO, Principal Investigator — Professor of NMM/OMM and Chief Medical Officer of WesternU Health
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No